CLINICAL TRIAL: NCT01838421
Title: Correlation of the Paediatric Tracheal Tube Size With the Known Formulas for the Calculation of the Size
Brief Title: Correlation of the Paediatric Tracheal Tube Size
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany
Other Study IDs: Paediatric tube size
Record Dates: First submitted 2013-04-02; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Pediatric Tracheal Tube Size

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children under 12 years of age: Children under 12 years of age who underwent surgery in the Charité - University Medicine Berlin, Campus Virchow - Klinikum in the years 2011/12

SUMMARY:
In the context of the study a retrospective data collection of all anaesthesia protocols of children under the age of 12 which underwent surgery in the Charité - University Medicine Berlin, Campus Virchow - Klinikum in the years 2011 and 2012 shall be executed. The correlation of the tracheal tube sizes with the weight, age and height shall be evaluated. This data collection should serve to reevaluate the already published formulas e.g. (Rettberg M. et al., 2011).

ELIGIBILITY:
Inclusion Criteria:

* Children under the age of 12 who underwent surgery in the Charité - University Medicine Berlin, Charité Campus Virchow - Klinikum in the years 2011/12

Exclusion Criteria:

* No endotracheal tube inserted

Ages: 1 Day to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under the age of 12 who underwent surgery in the Charité - University Medicine Berlin, Campus Virchow - Klinikum in the years 2011/12
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Correlation of the tracheal tube size with the known formulas for the calculation of the size. Correlation of the tracheal tube size with the known formulas for the calculation of the size | 24 month data capture
  For many years different weight, height, and/or age-based formulas have been published. The aim of the present study was to identify and to compare published formulas to estimate optimal tube size in pediatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Chair — Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] von Rettberg M, Thil E, Genzwurker H, Gernoth C, Hinkelbein J. [Endotracheal tubes in pediatric patients. Published formulas to estimate the optimal size]. Anaesthesist. 2011 Apr;60(4):334-42. doi: 10.1007/s00101-010-1756-0. German. PMID 20593158